CLINICAL TRIAL: NCT06414967
Title: Pilot Study Evaluating the Benefits of Music Therapy Combined With Conventional Treatment on Irritability and Impulsivity in Patients With Huntington's Disease (MUSIC-HD)
Brief Title: Study to Evaluate Music Therapy on Irritability and Impulsivity in Patients With Huntington's Disease (MUSIC-HD)
Acronym: MUSIC-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSIC-HD
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Huntington Disease
Keywords: Music Therapy; Irritability; Impulsivity
MeSH Terms: conditions — Huntington Disease; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Intervention (Experimental): The rythm of the music sessions will be 1 per week in the first month and every 15 days in the second and third month.
  Interventions: Other: Music Intervention

INTERVENTIONS:
Other: Music Intervention — Music therapy carried out with Music Care

SUMMARY:
The study is an open-label clinical trial evaluating whether music therapy combined with conventional management reduces irritability and impulsivity in 15 patients with early-stage Huntington's disease. This pilot study aims to show the interest of alternative non-pharmacological measures such as a digital music therapy tool, adapted to an audience of Huntington's patients, to help manage the psychobehavioral symptoms frequently observed in this affection, and to avoid breakdowns due to caregiver exhaustion.

DETAILED DESCRIPTION:
The participants will be recruited at the Clinical Investigation Center (CIC) of the University Hospital of Poitiers and will receive music therapy for 3 months.

After the start of the musical intervention, 3 visits (at 1 month, 3 months and 6 months) will be performed by practitioners, nurses and neuropsychologist at the CIC. Participants will answer questionnaires : irritability (BITe and PBA-s sub-score), impulsivity (UPPS-P and Delay discounting task), anxiety (STAI-Y and HAM-A), and quality of life: H-QoL-I. Caregivers will be asked to rate the patient's irritability and anxiety using a Lickert scale from 0 to 10, and the patient's impulsivity with the ISDC.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Huntington disease genetically confirmed by the presence of at least 35 repeats of the CAG triplet in exon 1 of the HTT gene
* UHDRS (Unified Huntington's disease Rating Scale) score <= 5 with a diagnostic confidence score =4
* Absence of significant cognitive impairment MoCA >=24
* Stable drug therapy in the 28 days prior inclusion and during the study
* Without legal tutors or subordination
* Affiliated to a health insurance system as required by the French law on biomedical research
* Written informed consent for participation in the study

Exclusion Criteria:

* Inability to give free and informed consent for study participation
* Significant hearing impairment
* Participating to another study the day of enrollement
* Persons benefiting from enhanced protection, i.e.persons deprived of their liberty by a judicial or administrative decision, adults under legal and finally patients in a vital emergency situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Describe evolution of irritability in patients with Huntington's disease after 3 months of music therapy combined with conventional management | Month 3
  Score of The brief Irritability Test (BITe). It consists of 5 questions, each rated on likert-type scale with 6 responses options, each question scores to 1 to 6. Lower score means a better outcome.

SECONDARY OUTCOMES:
Describe evolution of irritability in patients with Huntington's disease with music therapy combined with conventional management | Month [1;3;6]
  Score of The brief Irritability Test (BITe). It consists of 5 questions, each rated on likert-type scale with 1-6 responses options. Lower score means a better outcome.
  Score of Problem Behavior Assessment-short version (PBA-s). It consist of 4 questions, each rated on likert-type scale with 5 responses options, each question scores to 0 to 4. Lower score means a better outcome.
Describe evolution of impulsivity | Month [1;3;6]
  UPPS (Impulsive Behavior Scale). It consists of 20 questions, each rated on likert-type scale with 4 response options. Lower scores mean a better outcome.
  Delay discounting task. ISDC (Inventary of Comportement Dyexecutif Syndrom). It consists of 8 questions, each rated on likert-type scale with 3-5 response options. Lower scores means a better outcome.
Describe evolution of Anxiety. | Month [1;3;6]
  STAI-Y (Form-Y of the State-Trait Anxiety Inventory) score. It consist of 20-item scales providing separate measures of state and trait anxiety (S-Anxiety and T-Anxiety, respectively). On a 4-point Likert scale (1-4), a score equal to 4 indicates the presence of a higher level of anxiety.
  HAM-A (Hamilton Anxiety Rating Scale) score. It consist of 14 item-scale, each rated on likert-type scale with 4 response options. Lower scores mean a better outcome
Describe evolution of the quality of life | Month [3;6]
  H-QoL-I (Huntington Qualty of Life Instrument), It consist of 11 items scale, each rated on likert-type scale with 5 response options.Lower scores mean a better outcome.
Compliance with musical sessions | Month [1;3]
  Number of music therapy sessions performed.
Describe caregivers feeling about the effect of music intervention on patient's irritability and anxiety | Month [3;6]
  A lickert scale from 0 to 10. Lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers / CIC, Poitiers, France